CLINICAL TRIAL: NCT04376177
Title: Evaluation Des Mesures Dopplers, Angiographiques, Radiographique Oximetriques, Plethysmographiques, Electromyographiques et Des Questionnaires Cliniques Des Patients adressés Pour Suspicion de Syndrome du défilé Thoraco-brachial
Brief Title: Clinical Routine in Thoracic Outlet Syndrome
Acronym: SKIPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/17
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Ultrasonography; Angiography; Blood Gas Monitoring, Transcutaneous; Plethysmography; Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Thoracic outlet syndrome: Patients referred to the University Hospital of Angers for the diagnostis or follow-up of thoracic outlet syndrome
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: angiography; Diagnostic Test: questionnaires; Diagnostic Test: Transcutaneous oximetry; Diagnostic Test: plethysmography; Diagnostic Test: Electromyogram; Diagnostic Test: Standard X-Ray

INTERVENTIONS:
Diagnostic Test: Ultrasound — Echodoppler imaging of upper limbs performed by trained operators at rest and during provocative maneuvers for TOS diagnosis.
Diagnostic Test: angiography — Angiography (arterial and/or venous) of upper limbs performed by trained operators at rest and during provocative maneuvers such for TOS diagnosis.
Diagnostic Test: questionnaires — Use of standard questionnaires (MASC, DASH, SF36) for the evaluation of upper limb symptoms self-completed by the patients at admission.
Diagnostic Test: Transcutaneous oximetry — Mesurement of transcutaneuos oxygen pressure on both forearms performed at rest and during provocative maneuversfor TOS diagnosis.
Diagnostic Test: plethysmography — Photoplethysmography of the forearms or fingers performed at rest and during provocative maneuvers for TOS diagnosis
Diagnostic Test: Electromyogram — Electromyography of the upper limbs with encoding of the physician for the presence or abnsence of signs of plexis compression (impairment of the response on C8 T1 erea
Diagnostic Test: Standard X-Ray — Standard X-Ray performed for the research of apophysomegaly or additionnal cervical rib.

SUMMARY:
Transversal recording and analysis of investigations performed in patients referred for suspected thoracic outlet syndrome (TOS)

DETAILED DESCRIPTION:
Patients will have recording on a database of all investigations that were eventually performed for the diagnosis or follow up of their disease, among which:

* Characteristics (Age, Gender height, weight, ongoing treatment ,
* professional activity, sports activity,
* Symptoms.
* Forearm and finger photoplethysmography (PPG) during provocative maneuvers of the upper limb
* Transcutaneous oxymetry (Tcpo2) recording
* Standard questionnaires (MASC, DASH, FS36)
* Doppler and ultrasound during provocative maneuvers of the upper limb
* Angiography during provocative maneuvers of the upper limb
* Electromyogram
* Standard X-ray

ELIGIBILITY:
Inclusion Criteria:

* Absence of deny for the use of medical filesfor research purposes

Exclusion Criteria:

* Inability to understand the purpose of the database.
* Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult subjects referred for the diagnosis or follow up of TOS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ultrasound | 1 hour
  Retrieval of ultrasound interpretation as recorded in the patients' file by the physician that performed the test

OTHER OUTCOMES:
angiography encoding | 1 week
  Retrieval of angiography interpretation as recorded in the patients' file by the physician that performed the test
Questionnaire scoring | 1 hour
  Scoring of the questionnaires according to their respective scoring methods
Transcutaneous oximetry | 1 hour
  Recording of the decrease from rest of oxygen pressure (DROP) minimal value observed during the provocative maneuvers
Plethysmography interpretation | 1 hour
  Analysis of the pattern of volume changes observed during provocative maneuvers

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University and univerity hospital in Angers, FRANCE
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Hersant J, Lecoq S, Ramondou P, Feuilloy M, Abraham P, Henni S. Upper arm versus forearm transcutaneous oximetry during upper limb abduction in patients with suspected thoracic outlet syndrome. Front Physiol. 2022 Nov 8;13:1033137. doi: 10.3389/fphys.2022.1033137. eCollection 2022. PMID 36425296
- [Derived] Hersant J, Ramondou P, Josse C, Lecoq S, Henni S, Abraham P. Quantitative analysis of venous outflow with photo-plethysmography in patients with suspected thoracic outlet syndrome. Front Cardiovasc Med. 2022 Oct 28;9:803919. doi: 10.3389/fcvm.2022.803919. eCollection 2022. PMID 36386307